CLINICAL TRIAL: NCT03763942
Title: Theoretically Based Mobile App to Increase PrEP Uptake Among MSM
Brief Title: HealthMindr App to Increase Pre-exposure Prophylaxis (PrEP) Uptake and Retention Among Men Who Have Sex With Men (MSM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Patrick S Sullivan, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00102006; R01DA045612 (NIH)
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Results first posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: HIV Infections
Keywords: Human Immunodeficiency Virus (HIV); Men who have sex with men (MSM); Pre-Exposure Prophylaxis (PrEP); HealthMindr
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Homosexuality

STUDY DESIGN:
Intervention Model Description: This trial will include 657 participants with 2:1 allocation for the intervention (438) and control (219) conditions. Recruitment strategies will be formulated to increase enrollment of MSM who identify as members of racial/ethnic minority groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HealthMindr App (Experimental): Participants in the intervention arm will receive access to all HealthMindr app capabilities. The app information will cover the importance of testing, links to HIV prevention resources, resources to locate HIV testing and PrEP services, the Substance Abuse and Mental Health Services Administration (SAMHSA) substance abuse treatment resource locator, and other prevention information specific to their area.
  Interventions: Behavioral: HealthMindr App
- Control App (Placebo Comparator): Participants in the control arm will be directed to download a study app that allows study staff to interact with them.
  Interventions: Behavioral: Control App

INTERVENTIONS:
Behavioral: HealthMindr App — Participants in the intervention arm will receive access to the HealthMindr app with basic prevention services (HIV test planning and test locators; risk assessment; HIV treatment locators; and condom, HIV test kit, and at-home STI specimen collection kit distribution) plus monthly PrEP eligibility assessments, PrEP provider locator, enhanced information about PrEP, and referrals to local PrEP navigators. The app also provides information about obtaining health insurance coverage and paying for PrEP.
  Arms: HealthMindr App
Behavioral: Control App — Men in the control arm will have access to an app with information pertinent to their participation in the study, including a study events timeline. The app will also allow participants and study staff to communicate via a messaging feature. The control arm app will not contain HIV prevention information.
  Arms: Control App

SUMMARY:
This study is a randomized controlled clinical trial of a theoretically based mobile app, HealthMindr, to increase pre-exposure prophylaxis (PrEP) uptake among men who have sex with men (MSM) to prevent human immunodeficiency virus (HIV). Participants in the intervention arm will receive access to the HealthMindr app, with information about PrEP and other HIV prevention methods in addition to provider locators. Participants randomized to the control arm will receive standard of care. The primary aim for this study is to assess PrEP uptake in the intervention arm compared to the control arm.

DETAILED DESCRIPTION:
MSM are disproportionately impacted in terms of HIV prevalence and incidence. Electronically delivered or supported prevention services are effective, are acceptable to MSM, and will likely reach heavily impacted men. The study is based on the premise that providing, through a mobile phone app, self-directed PrEP information; periodic behavioral screenings to identify HIV risk and PrEP indication objectively; referral to PrEP providers with directions; and related prevention services will increase the uptake of PrEP among at risk, HIV negative MSM to a greater extent than standard of care referrals to existing resources.

The study will examine the effectiveness of the HealthMindr app to increase uptake of PrEP among MSM. The study will enroll 657 men across the three sites - the metropolitan statistical areas (MSA) of Atlanta, Georgia (GA), Jackson, Mississippi (MS), and Washington, D.C. - into a randomized controlled trial. Participants in the intervention arm will receive access to the HealthMindr app and men in the control arm will receive standard of care HIV prevention information. PrEP uptake will be assessed during follow-up by self-report at months 3, 6, 9, and 12. Self-report will be confirmed by laboratory testing for the presence of tenofovir diphosphate (TFV-DP) and/or photograph of PrEP prescription or bottle.

At the beginning of the study, all participants will download a study mobile app. After completing a baseline survey, participants will be randomized to the intervention or control arm. For participants assigned to the intervention arm, additional app content will become available. This content will include information about basic prevention services (HIV test planning and test locators; risk assessment; HIV treatment locators; and condom, HIV test kit, and at-home sexually transmitted infection (STI) specimen collection kit distribution) plus monthly PrEP eligibility assessments, PrEP provider locator, enhanced information about PrEP, and referrals to local PrEP navigators. The app also provides links to health insurance exchanges, where men can seek health insurance or assistance to help cover PrEP costs. The control arm will be referred to existing online PrEP and HIV prevention information. Participants in the control arm will access the control version of the app that contains elements pertinent to their participation in the research study.

Additional follow-up surveys will be conducted at 3, 6, 9, and 12 months and participants will also complete monthly assessments. The monthly assessments will assess indications for PrEP and PrEP uptake (intervention arm) and other health-related behaviors (control arm). Participants reporting PrEP initiation will be asked to submit a dried blood spot self-collection kit to allow for measurement of tenofovir diphosphate (TFV-DP) levels and/or upload a photo of their PrEP prescription bottle to verify PrEP uptake.

Participants will primarily be recruited online from the main study sites in Atlanta, Georgia, Jackson, Mississippi, and Washington, District of Columbia (DC). Online recruitment will expand to other areas of the United States, as needed to meet recruitment targets.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender male
* 18-34 years of age (inclusive)
* Resides in one of the study MSAs
* Intends to remain in study area for duration of the trial
* Owns an Android or Apple operating system (iOS) smartphone and willing to download study app
* Able to read and understand English without assistance
* Reports having anal sex with a man in the past 6 months
* Reports being HIV negative or never tested for HIV

Exclusion Criteria:

* Cisgender female, transgender male, transgender female, gender non-conforming
* Currently on PrEP
* < 18 or >34 years of age
* Reports being HIV positive
* Resides outside of the MSAs or plans to move outside study MSA within 12 months
* Current participant in another HIV prevention study
* Unable to download study app

Ages: 18 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 658 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Sullivan, DVM PhD, Principal Investigator — Emory University; Jeb Jones, PhD, Study Director — Emory University
Locations (3):
- United States (3):
  - George Washington University, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - University of Mississippi Medical Center, Jackson, Mississippi

REFERENCES:
- [Background] Jones J, Dominguez K, Stephenson R, Stekler JD, Castel AD, Mena LA, Jenness SM, Siegler AJ, Sullivan PS. A Theoretically Based Mobile App to Increase Pre-Exposure Prophylaxis Uptake Among Men Who Have Sex With Men: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Feb 21;9(2):e16231. doi: 10.2196/16231. PMID 32130178

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The following report is based on 658 consented participants that took part in the study.
Period: Overall Study
Arm/Group | HealthMindr App | Control App
Started | 437 | 221
Completed | 318 | 164
Not Completed | 119 | 57
Not completed — Lost to Follow-up | 114 | 54
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Other | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HealthMindr App | Control App | Total
Number analyzed (Participants) | 437 | 221 | 658
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.83 (4.23) | 27.08 (4.47) | 26.91 (4.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 437 | 221 | 658
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 100 | 52 | 152
  Not Hispanic or Latino | 337 | 169 | 506
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 437 | 221 | 658
Household Income [Count of Participants; unit: Participants] — Population: Discrepancies in number of participants analyzed are due to missing data for one participant in each study group.
  Participants
    $0-29,999/year: number analyzed (Participants) | 436 | 220 | 656
    $0-29,999/year | 135 | 75 | 210
    $30,000-74,999/year: number analyzed (Participants) | 436 | 220 | 656
    $30,000-74,999/year | 187 | 91 | 278
    $75,000+: number analyzed (Participants) | 436 | 220 | 656
    $75,000+ | 91 | 42 | 133
    Unknown: number analyzed (Participants) | 436 | 220 | 656
    Unknown | 23 | 12 | 35
Educational Status [Count of Participants; unit: Participants]
  High school or less | 42 | 22 | 64
  Less than 4 years of college (Includes technical or vocational school) | 96 | 48 | 144
  4-year college grad or higher | 299 | 151 | 450
Employment status [Count of Participants; unit: Participants] — Population: Discrepancy in total number of patients analyzed is due to missing data for one participant in the HealthMindr App Group.
  Participants
    Not currently employed: number analyzed (Participants) | 436 | 221 | 657
    Not currently employed | 82 | 47 | 129
    Employed full time: number analyzed (Participants) | 436 | 221 | 657
    Employed full time | 288 | 129 | 417
    Employed part time: number analyzed (Participants) | 436 | 221 | 657
    Employed part time | 66 | 45 | 111
Health Insurance Status [Count of Participants; unit: Participants]
  Private | 303 | 143 | 446
  Public | 41 | 19 | 60
  Other/Don't know | 8 | 8 | 16
  No insurance | 85 | 51 | 136
Housing [Count of Participants; unit: Participants] — Population: Discrepancies in number of participants analyzed are due to missing data for two participants in each study group.
  Participants
    Stable/permanent: number analyzed (Participants) | 435 | 219 | 654
    Stable/permanent | 358 | 174 | 532
    Transitional/temporary: number analyzed (Participants) | 435 | 219 | 654
    Transitional/temporary | 68 | 39 | 107
    Homeless: number analyzed (Participants) | 435 | 219 | 654
    Homeless | 7 | 4 | 11
    Other: number analyzed (Participants) | 435 | 219 | 654
    Other | 1 | 0 | 1
    Unknown: number analyzed (Participants) | 435 | 219 | 654
    Unknown | 1 | 2 | 3
Food Insecurity [Count of Participants; unit: Participants] — Food insecurity was assessed using the following question:
  In the past 12 months, did you or other adults in the household ever cut the size of your meals or skip meals because there wasn't enough money for food?
  Number of responses were counted for the answers:
  "Yes", "No","Don't know" and "Prefer not to answer". Population: Discrepancies in number of participants analyzed are due to missing data for 4 participants in the Control App group.
  Participants
    Yes: number analyzed (Participants) | 437 | 217 | 654
    Yes | 83 | 48 | 131
    No: number analyzed (Participants) | 437 | 217 | 654
    No | 343 | 162 | 505
    Unknown: number analyzed (Participants) | 437 | 217 | 654
    Unknown | 2 | 3 | 5
    Prefer not to answer: number analyzed (Participants) | 437 | 217 | 654
    Prefer not to answer | 9 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: PrEP Uptake
Description: PrEP uptake was assessed at each follow-up timepoint (3, 6, 9, and 12 months) in the intervention and control groups. The primary measure of PrEP uptake will be self-report. Validation will occur through submission of a dried blood spot self-collection kit to detect tenofovir diphosphate (TFV-DP) and/or upload of a photo of a PrEP prescription bottle.
Time Frame: 3, 6, 9, and 12 months post-randomization
Population: Number of participants analyzed per different time point are based on number of patient that were able to complete the corresponding study visit.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-months
Arm/Group | HealthMindr App | Control App
Number analyzed (Participants) | 358 | 190
events per 1000 person-months
  PrEP Uptake at 3 months post-randomization | 2.764 [2.211 to 3.414] | 2.116 [1.482 to 2.929]
  PrEP Uptake at 6 months post-randomization: number analyzed (Participants) | 334 | 178
  PrEP Uptake at 6 months post-randomization | 2.104 [1.737 to 2.525] | 1.837 [1.384 to 2.391]
  PrEP Uptake at 9 months post-randomization: number analyzed (Participants) | 325 | 163
  PrEP Uptake at 9 months post-randomization | 1.762 [1.477 to 2.085] | 1.509 [1.157 to 1.935]
  PrEP Uptake at 12 months post-randomization: number analyzed (Participants) | 318 | 164
  PrEP Uptake at 12 months post-randomization | 1.241 [1.033 to 1.480] | 1.462 [1.146 to 1.838]

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the baseline assessment and continued through the final assessment at 12 months post-intervention.
Arm/Group | HealthMindr App | Control App
All-Cause Mortality (participants affected / at risk) | 0/437 | 0/221
Serious Adverse Events (participants affected / at risk) | 0/437 | 0/221
Other Adverse Events (participants affected / at risk) | 0/437 | 0/221

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT03763942/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT03763942/ICF_000.pdf